CLINICAL TRIAL: NCT01711554
Title: A Phase I Study of Lenalidomide and Anti-GD2 Mab Ch14.18 +/- Isotretinoin in Patients With Refractory/Recurrent Neuroblastoma
Brief Title: Lenalidomide and Dinutuximab With or Without Isotretinoin in Treating Younger Patients With Refractory or Recurrent Neuroblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02011; NCI-2012-02011 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000741991; N2011-04; NANT 11-04; NANT N2011-04 (Other: New Approaches to Neuroblastoma Therapy (NANT)); NANT N2011-04 (Other: CTEP); P01CA081403 (NIH)
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Neuroblastoma; Refractory Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — dinutuximab; Isotretinoin; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (lenalidomide, dinutuximab, isotretinoin) (Experimental): Patients receive lenalidomide PO QD on days 1-21, dinutuximab IV over 10 hours on days 8-11, and isotretinoin PO BID on days 15-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Dinutuximab; Drug: Isotretinoin; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Other: Pharmacological Study

INTERVENTIONS:
Biological: Dinutuximab — Given IV
  Other Names: Ch 14.18UTC; Ch14.18; Dinutuximab Beta; MOAB Ch14.18; monoclonal antibody Ch14.18; Qarziba; Unituxin
Drug: Isotretinoin — Given PO
  Other Names: 13-cis retinoic acid; 13-cis-Retinoate; 13-cis-Retinoic Acid; 13-cis-Vitamin A Acid; 13-cRA; Absorica; Accure; Accutane; Amnesteem; cis-Retinoic Acid; Cistane; Claravis; Isotretinoinum; Isotrex; Isotrexin; Myorisan; Neovitamin A; Neovitamin A Acid; Oratane; Retinoicacid-13-cis; Ro 4-3780; Ro-4-3780; Roaccutan; Roaccutane; Roacutan; Sotret; ZENATANE
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of lenalidomide when given together with dinutuximab with or without isotretinoin in treating younger patients with neuroblastoma that does not respond to treatment or that has come back. Drugs used in chemotherapy, such as lenalidomide and isotretinoin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as dinutuximab, may interfere with the ability of tumor cells to grow and spread. Giving more than one drug (combination chemotherapy) together with dinutuximab therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) of lenalidomide in combination with fixed doses of dinutuximab (ch14.18) and isotretinoin given to children with refractory or recurrent neuroblastoma.

II. To define the toxicities of lenalidomide administered in combination with ch14.18 and isotretinoin.

III. To describe the differences in immune function modulation between "low" versus "high" dose lenalidomide given with ch14.18 and isotretinoin.

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetics of lenalidomide given in this combination regimen.

II. To determine the steady state pharmacokinetics of isotretinoin (day 28, course one) given in combination with lenalidomide.

III. To measure peak and trough levels of ch14.18 in patients receiving lenalidomide and to compare to historical controls of patients receiving ch14.18 in combination with interleukin 2 (IL-2) and granulocyte-macrophage colony-stimulating factor (GM-CSF).

IV. To describe the immunological effects of lenalidomide (T cells, natural killer [NK] cells, monocytes, cytokines, chemokines) within this three drug regimen.

V. To define the incidence and titers of human anti-chimeric antibody (HACA) on this regimen.

VI. To describe, within the context of a phase I study, the response rate to lenalidomide combined with ch14.18 and isotretinoin in patients with recurrent/refractory neuroblastoma.

VII. To summarize, within the context of a phase I study, the event-free survival of patients with recurrent/refractory neuroblastoma or in complete response (CR) after progressing, and who are treated with lenalidomide combined with ch14.18 and isotretinoin.

VIII. To determine, within the context of a phase I study, if killer-cell immunoglobulin-like receptor (KIR) receptor-ligand mismatch or specific Fc gamma receptor (Fc gamma R) alleles are associated with anti-tumor response.

IX. To quantify neuroblastoma tumor cell "load" using a 5-gene TaqMan Low Density Array (TLDA) assay in peripheral blood at study entry, following, with each disease evaluation and at end of therapy and bone marrow at study entry, with each response evaluation when bone marrow is sampled, and at end of therapy.

X. To compare the toxicities of this regimen with the historical toxicity data from the Children's Oncology Group (COG) ANBL0032 and ANBL0931 studies of ch14.18 with IL-2, GM-CSF and isotretinoin.

XI. To describe the tolerability and ability to give full doses of ch14.18 and lenalidomide over extended periods of time, i.e. in courses 6-12.

OUTLINE: This is a dose-escalation study of lenalidomide.

Patients receive lenalidomide orally (PO) once daily (QD) on days 1-21, dinutuximab intravenously (IV) over 10 hours on days 8-11, and isotretinoin PO twice daily (BID) on days 15-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of neuroblastoma either by histologic verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines
* Patients must have high-risk neuroblastoma
* Patients must have at least ONE of the following:

  * Recurrent/progressive disease at any time prior to enrollment - regardless of response to frontline therapy
  * Refractory disease: persistent sites of disease (after less than a partial response to frontline therapy, following a minimum of 4 cycles of induction therapy) AND patient has never had a relapse/progression
  * Persistent disease: persistent disease after achieving at least a partial response to frontline therapy after a minimum of 4 cycles of induction therapy and patient has never had a relapse/progression
* Patients must have at least ONE of the following (lesions may have received prior radiation therapy as long as they meet the other criteria listed below):

  * Bone disease

    * At least one metaiodobenzylguanidine (MIBG) avid bone site or diffuse MIBG uptake

      * For recurrent/progressive or refractory disease a biopsy is not required regardless of number of MIBG avid lesions
      * For persistent disease, if patient has only 1 or 2 MIBG avid lesions OR a Curie score of 1-2, then biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma in at least one site present at the time of enrollment (bone marrow, bone, or soft tissue) is required to be obtained at any time point prior to enrollment and two weeks subsequent to most recent prior therapy; if a patient has 3 or more MIBG avid lesions OR a Curie score of >= 3 then no biopsy is required for eligibility
    * If a tumor is known to be MIBG non-avid, then a patient must have at least one fludeoxyglucose (FDG)-positron emission tomography (PET) avid bone site present at the time of enrollment with biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma obtained at any time prior to enrollment and two weeks subsequent to most recent prior therapy
  * Any amount of neuroblastoma tumor cells in the bone marrow based on routine morphology (with or without immunocytochemistry) in at least one sample from bilateral aspirates and biopsies
  * At least one soft tissue lesion that meets the criteria for a TARGET lesion as defined by:

    * SIZE: Lesion can be accurately measured in at least one dimension with a longest diameter >= 10 mm, or for lymph nodes >= 15 mm on short axis; lesions meeting size criteria will be considered measurable
    * In addition to size, a lesion needs to meet ONE of the following criteria:

      * MIBG avid; for patients with persistent disease only: if a patient has only 1 or 2 MIBG avid lesions OR a Curie score of 1-2, then biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma in at least one site present at time of enrollment (either bone marrow, bone and/or soft tissue) is required to be obtained at any time point prior to enrollment and at least two weeks subsequent to most recent prior therapy; if a patient has 3 or more MIBG avid lesions OR a Curie score of >= 3 then no biopsy is required for eligibility
      * FDG-PET avid (only if tumor is known to be MIBG non-avid); these patients must have had a biopsy confirming neuroblastoma and/or ganglioneuroblastoma in at least one FDG-PET avid site present at the time of enrollment done prior to enrollment and at least two weeks subsequent to the most recent prior therapy
      * Non-avid lesion (both MIBG and FDG-PET non-avid); these patients must have had a biopsy confirming neuroblastoma and/or ganglioneuroblastoma in at least one non-avid lesion present at the time of enrollment done prior to enrollment and at least two weeks subsequent to the most recent prior therapy
* Patients with prior progressive disease who do not meet criteria above, are eligible as long as they have not been off treatment for > 3 months prior to enrollment on NANT 2011-04
* Patients must have a life expectancy of at least 6 weeks
* Lansky (=< 16 years) or Karnofsky (> 16 years) score of at least 50
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to study enrollment
* Patients must not have received the therapies indicated below for the specified time period prior to the first day of administration of protocol therapy on this study

  * Myelosuppressive chemotherapy: must have received last dose at least 2 weeks prior to protocol therapy; this includes cytotoxic agents given on a low dose metronomic regimen
  * Biologic (anti-neoplastic agent) (includes retinoids): must have received last dose at least 7 days prior to protocol therapy
  * Monoclonal antibodies: must have received last dose at least 7 days or 3 half-lives, whichever is longer, prior to protocol therapy
* Radiation:

  * Patients must not have received radiation (small port) for a minimum of two weeks prior to protocol therapy
  * Except for patients with a history of progressive disease, patients whose only site(s) of disease have been radiated are eligible if at least one lesion meets at least one of the criteria listed in sites of disease above
  * A minimum of 12 weeks prior to start of protocol therapy is required following large field radiation therapy (i.e. total body irradiation, craniospinal, whole abdominal, total lung, > 50% marrow space)
  * A minimum of 6 weeks must have elapsed prior to start of protocol therapy for other substantial bone marrow radiation
* Stem Cell Transplant (SCT):

  * Patients are eligible 6 weeks after date of autologous stem cell infusion following myeloablative therapy (timed from first day of protocol therapy)
  * Patients are not eligible post allogeneic stem cell transplant
  * Patients who have received an autologous stem cell infusion to support non-myeloablative therapy (such as 131 iodine [I]-MIBG) are eligible at any time as long as they meet the other criteria for eligibility
* A minimum of 6 weeks must have elapsed after 131I-MIBG therapy prior to start of protocol therapy
* Prior anti-disialoganglioside (GD2) antibody, isotretinoin, or lenalidomide therapy:

  * Patients who have received prior anti-GD2 antibody therapy are eligible if they did not have tumor relapse/progression while receiving this therapy
  * Patients who have received either isotretinoin or lenalidomide are eligible, but not if they have received the two agents concomitantly
* All cytokines or hematopoietic growth factors must be discontinued a minimum of 7 days prior to protocol therapy
* Patients must not be receiving any other anti-cancer agents or radiotherapy at the time of study entry or while on study
* Absolute phagocyte count (APC = neutrophils and monocytes): >= 1000/mm^3
* Absolute neutrophil count: >= 750/mm^3
* Platelet count: >= 50,000/mm^3, transfusion independent (no platelet transfusions within 1 week)
* Hemoglobin >= 8.0 (may transfuse)
* Patients with known bone marrow metastatic disease will be eligible for study as long as they meet hematologic function criteria; patients with marrow disease are not evaluable for hematologic toxicity
* Age-adjusted serum creatinine =< 1.5 x normal for age or creatinine clearance or glomerular filtration rate (GFR) >= 60 cc/min/1.73 m^2

  * Age 1 month to < 6 months: 0.4 mg/dL for males and 0.4 mg/dL for females
  * Age 6 months to < 1 year: 0.5 mg/dL for males and 0.5 mg/dL for females
  * Age 1 to < 2 years: 0.6 mg/dL for males and 0.6 mg/dL for females
  * Age 2 to < 6 years: 0.8 mg/dL for males and 0.8 mg/dL for females
  * Age 6 to < 10 years: 1.0 mg/dL for males and 1.0 mg/dL for females
  * Age 10 to < 13 years: 1.2 mg/dL for males and 1.2 mg/dL for females
  * Age 13 to < 16 years: 1.5 mg/dL for males and 1.4 mg/dL for females
  * Age >= 16 years: 1.7 mg/dL for males and 1.4 mg/dL for females
* =< grade 2 hematuria (criteria applicable only for dose levels that include isotretinoin) and =< grade 2 proteinuria
* Total bilirubin =< 1.5 x upper limit of normal for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 and serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 3 x upper limit of normal (note that for ALT, the upper limit of normal is defined as 45 U/L)
* Sinusoidal obstruction syndrome (SOS) if present, must be stable or improving clinically
* Cardiac function:

  * Normal ejection fraction (>= 55%) documented by either echocardiogram or radionuclide multi gated acquisition scan (MUGA) evaluation; OR
  * Normal fractional shortening (>= 27%) documented by echocardiogram
* No dyspnea at rest
* Serum triglyceride =< 300 mg/dL (applicable only for dose levels that include isotretinoin) (note that a non-fasting triglyceride value could be obtained, if this is > 300 mg/dL then a fasting triglyceride should be obtained and patient will be eligible if the fasting level is =< 300 mg/dL)
* =< grade 2 hypercalcemia (applicable only for dose levels that include cis retinoic acid [RA])
* Skin toxicity =< grade 1
* All post-menarchal females must have a negative beta-human chorionic gonadotropin (HCG); males and females of reproductive age and childbearing potential must use effective contraception for the duration of their participation; females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days and again within 24 hours prior to prescribing lenalidomide for cycle 1 and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy
* Patients with other ongoing serious medical issues must be approved by the study chair prior to registration

Exclusion Criteria:

* Quantitative serum b-HCG must be negative in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method; pregnant or breast-feeding women will not be entered on this study
* Breast feeding women are not eligible
* Patients who have an active or uncontrolled infection are excluded
* Patients with a paraben allergy cannot take isotretinoin preparations containing this compound (i.e. Accutane, Sotret) but are eligible if they can take an alternate preparation without paraben; (applicable only for entry onto dose levels receiving isotretinoin)
* Patients with a history of venous or arterial thrombosis personally before the age of 40 years unless associated with a central line
* Patients with a history of prior central nervous system (CNS) metastases or skull lesions with intracranial extension will be required to have a head computed tomography (CT) or magnetic resonance imaging (MRI) at study entry demonstrating no active CNS metastases; patients with skull metastases with associated intracranial soft tissue masses will remain eligible
* Inability to swallow lenalidomide capsules whole; capsules of 13-isotretinoin may be opened
* Patient declines participation in NANT 2004-05; unless the institution has been granted special exemption from mandatory enrollment on NANT 2004-05 by the NANT Operations Center

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2013-02-04 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2026-03-17 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose defined as the highest dose level tested at which 0/6 or 1/6 patients experience dose-limiting toxicity (DLT) graded using National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) criteria, version 4.0 | Up to 28 days
  All toxicities observed will be summarized in terms of type (organ affected or laboratory determination), severity (by NCI CTCAE), and attribution. Tables will be created to summarize these toxicities and side effects by dose level and by course as well as with Kaplan-Meier plots (i.e. time to first delay or dose reduction) in order to assess the tolerability of the regime over multiple courses.
Recommended phase II dose | Up to 28 days
  Determination of the recommended phase II dose of lenalidomide will include consideration of obtaining median peak plasma lenalidomide levels of 5-10 uM (based on laboratory modeling of this regimen in neuroblastoma), acceptable clinical toxicity, and laboratory evidence of an augmentation in immune function.

SECONDARY OUTCOMES:
Overall survival | From start of lenalidomide until death for any reason or date that patient was last known to be alive if the patient is still alive, assessed up to 3 years
  Will be summarized with Kaplan-Meier plots.
Event-free survival | From the start of treatment with lenalidomide until progression, clinical deterioration mandating that the patient terminate treatment or death due to any cause, whichever occurs first, assessed up to 3 years
  Will be summarized with Kaplan-Meier plots.
Changes in the levels of T cells, natural killer (NK) cells, monocytes, cytokines, and chemokines | Baseline to up to 28 days
  These levels and the changes relative to baseline will be summarized by dose level by simple summary statistics: means (possibly after transformation) or medians, ranges, and standard deviations (if numbers and distribution permit). Scatterplots will be used to explore possible associations between the dose and day and toxicity experienced (as reflected in the maximum grade of toxicity experienced, infections or platelet recovery).
Changes in levels of HACA (or other genotype) and tumor response | Baseline to up to 3 years
  These levels and the changes relative to baseline will be summarized by dose level by simple summary statistics: means (possibly after transformation) or medians, ranges, and standard deviations (if numbers and distribution permit). Scatterplots will be used to explore possible associations between the dose and day and toxicity experienced (as reflected in the maximum grade of toxicity experienced, infections or platelet recovery).
Pharmacokinetic determinations of lenalidomide | Baseline, at 60 and 90 minutes, at 2, 6, 24 hours and days 7 and 22 after last dose of lenalidomide in course 1
  These will be summarized by dose level with simple summary statistics: means (possibly after transformation) or medians, ranges, and standard deviations (if numbers and distribution permit). Scatterplots will be used to explore possible associations between the dose and estimates of the pharmacokinetic parameters, and between the pharmacokinetic determinations and toxicity experienced (as reflected in the maximum grade of toxicity experienced or in clinical measurements).
Changes in TaqMan low density array (TLDA) scores | Baseline to up to 3 years
  Standard descriptive summaries as well as scatterplots will be used. The association between the changes in TLDA scores and overall tumor response will also be summarized graphically and quantitatively. Changes (from baseline) in the TLDA scores over the course of treatment will be plotted and summarized by dose level and course.
Overall response | Up to 3 years
  The association between the changes in TLDA scores and overall tumor response will be summarized graphically and quantitatively.

CONTACTS AND LOCATIONS:
Overall Officials: Araz Marachelian, Principal Investigator — New Approaches to Neuroblastoma Treatment (NANT)
Locations (15):
- United States (14):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada